CLINICAL TRIAL: NCT03815799
Title: The Effect of Ultrasound-Guided Erector Spinae Block on Respiratory Function After Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya Meram State Hospital (Other)
Responsible Party: Principal Investigator, Asst. Prof. Munıse Yıldız M.D., Ass.Prof., Konya Meram State Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ESP-RF
Record Dates: First submitted 2019-01-04; First posted 2019-01-24 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Laparoscopic Cholecystectomy; Postoperative Pain; Respiratory Function
Keywords: Erector Spinae Block; Laparoscopy; Respiratory Function
MeSH Terms: conditions — Pain, Postoperative; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector Spinae Plane Block Group (Experimental): Procedure:
  In addition to routine standard perioperative and postoperative analgesic protocol participants will recieve erector spinae block under ultrasound guidence after the strict aseptic precautions.
  Interventions: Procedure: Bilateral Erector Spinae Block
- Control (Sham Comparator): Routine standard perioperative and postoperative analgesic protocol will be given.
  Interventions: Other: Control

INTERVENTIONS:
Procedure: Bilateral Erector Spinae Block — A linear ultrasound transducer will be place in a longitudinal parasagittal orientation about 3 cm lateral to spinous process. 40 ml bupivacaine/lidocaine mixture will be injected into the fascial plane on the deep aspect of erector spinae muscle. Standard perioperative and postoperative analgesia protocol will be given and postoperative pain levels will be determined by Numerical rating scale (NRS).
  Arms: Erector Spinae Plane Block Group
Other: Control — Standard perioperative and postoperative analgesia protocol will be given consisting of paracetamol 1 gr IV and tenoxicam 20 mg IV initiated after induction of anesthesia. At the end of the operation patients will receive meperidine 0.5 mg/kg IV before extubation. Postoperative pain levels will be determined by Numeric Rating Scale (NRS) system, 20 minutes intervals in the first hour and at 2th, 6th, 12th and 24 th hour. For the first hour in the postoperative care unit, tramadol 50 mg IV will be given for rescue analgesia with minimum 20 minutes between doses, in patients showing a NRS ≥ 4. Paracetamol 1 g / 12 hour will be given during ward follow-up. In the ward in patients showing a NRS ≥ 4 tramadol 50 mg IV will be given for analgesia.
  Arms: Control

SUMMARY:
The aim of this study is to assess the effect of ultrasound guided erector spinae block in control of the postoperative pain and the respiratory functions after laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

• American Society of Anesthesiology (ASA) physical status I-II patients who were scheduled for elective laparoscopic cholecystectomy

Exclusion Criteria:

* Patients refusal
* Contraindications for regional anesthesia
* Alcohol or drug abuse
* Chronic opioid intake
* Patient with psychiatric disorders
* Use of pain killers within the 24 h before the operation
* Respiratory tract infection within the last 2 weeks
* Smoker or history of smoking
* Allergy to local anesthetics
* Respiratory and allergic diseases
* Cardiac disease associated with dyspnea

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-03-03 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Scoring of postoperative pain | Postoperative 24 hour
  The primary outcome variable is Numeric Rating Scale (NRS) pain scores changes both at rest and movement. NRS use numbers to rate pain from 0 (no pain) to 10 (worst pain).

SECONDARY OUTCOMES:
Analgesic consumption | Postoperative 24 hour
  Total opioid consumption after the operation
Spirometric Parameters of Respiratory Functions | Preoperative (before the surgery) and at postoperative 24th hour
  Respiratory functions assessed by spirometric parameters (FEV1, FVC, FEV1/FVC, and PEFR)
Number of Adverse events | Postoperative 24 hour
  Postoperative nausea and vomiting incidents at PACU and and at ward.

CONTACTS AND LOCATIONS:
Locations (1):
- Konya Education and Training Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tulgar S, Kapakli MS, Senturk O, Selvi O, Serifsoy TE, Ozer Z. Evaluation of ultrasound-guided erector spinae plane block for postoperative analgesia in laparoscopic cholecystectomy: A prospective, randomized, controlled clinical trial. J Clin Anesth. 2018 Sep;49:101-106. doi: 10.1016/j.jclinane.2018.06.019. Epub 2018 Jun 15. PMID 29913392
- [Background] Basaran B, Basaran A, Kozanhan B, Kasdogan E, Eryilmaz MA, Ozmen S. Analgesia and respiratory function after laparoscopic cholecystectomy in patients receiving ultrasound-guided bilateral oblique subcostal transversus abdominis plane block: a randomized double-blind study. Med Sci Monit. 2015 May 7;21:1304-12. doi: 10.12659/MSM.893593. PMID 25948166
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016